CLINICAL TRIAL: NCT05238168
Title: ePIPARI - Digital Follow-up of Preterm Infants During First Two Years
Brief Title: Evaluation of Digital Follow up of Preterm Infants
Acronym: ePIPARI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other); University of Helsinki (Other)
Responsible Party: Principal Investigator, Liisa Lehtonen, Professor, Turku University Hospital
Other Study IDs: T200/2018
Record Dates: First submitted 2022-02-03; First posted 2022-02-14 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Preterm Birth; Development Delay; Sensory Disorder; Growth Disorders; Family Relations
Keywords: Preterm infant; Digital follow up; Electronic health monitoring
MeSH Terms: conditions — Premature Birth; Learning Disabilities; Sensation Disorders; Growth Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ePIPARI digital follow up tool — A digital platform includes questions to parents about child wellbeing and development and parent wellbeing. A notification by email or app comes two weeks before the follow up time point. The parents respond via a link to a webpage or via an app.They also receive information (text and video) about age-appropriate child development. ePIPARI includes 8 assessment points from term age until 2 years of corrected age.

SUMMARY:
The aim is to study how a digital follow up tool can identify the preterm born children and their families who need further support or clinical interventions

DETAILED DESCRIPTION:
This study runs a digital follow up parallel to clinical follow up, up to 2 years of corrected age of the child. It evaluates the ability of the digital follow up tool to identify the problems in growth and health, eating and feeding, neurodevelopment and parental wellbeing which require further support or interventions. This study includes all infants born under 34 weeks of gestation in Turku University Hospital during years 2019-2022 and those preterm children born under 32 weeks of gestation who turn to 2 years during years 2019-2021.

Parent satisfaction about the digital follow up tool is asked at each time point and anonymously once per year. The follow up age points are the expected day of birth, 1 month, 2 months, 4 months, 8 months, 12 months, 18 months and 24 months after the expected birth date.

ELIGIBILITY:
Inclusion Criteria:

* Children born before 34 weeks fo gestation and their parents
* Clinical follow up at Turku University Hospital

Exclusion Criteria:

* Parents do not speak Finnish, Swedish or English

Ages: 1 Month to 28 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants treated in a neonatal intensive care unit and their parents.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Ability to identify children and parents in need for further support/interventions questionnaire | 0-28 months
  Digital follow up tool is compared to clinical follow up
Response rate | 0-28 months
  How many families responded at each time point

SECONDARY OUTCOMES:
Parent satisfaction Questionnaire | 0-28 months
  Questionnaire at each time point after the digital follow up and anonymous once yearly

CONTACTS AND LOCATIONS:
Overall Officials: Liisa Lehtonen, MD, Principal Investigator — Turku University Hospital
Locations (1):
- NICU/Pediatrics, Turku, Finland

REFERENCES:
- [Derived] Saarinen T, Ylijoki M, Lehtonen L, Munck P, Stolt S, Lapinleimu H, Rautava P, Haataja L, Setanen S, Leppanen M, Huhtala M, Saarinen K, Gronroos L, Korja R; PIPARI Study group. Web-based follow-up tool (ePIPARI) of preterm infants-study protocol for feasibility and performance. BMC Pediatr. 2023 Aug 23;23(1):413. doi: 10.1186/s12887-023-04226-4. PMID 37612695